CLINICAL TRIAL: NCT01537575
Title: Intravenous Immunoglobulins for Post-Polio Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Laura Bertolasi, Head of the Neurophysiology Unit, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUDRACT-200700-3559-35
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Post-polio Syndrome
MeSH Terms: conditions — Postpoliomyelitis Syndrome | interventions — Immunoglobulins, Intravenous; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline solution (Placebo Comparator)
  Interventions: Biological: Saline solution
- intravenous immunoglobulins (Experimental)
  Interventions: Biological: intravenous immunoglobulins

INTERVENTIONS:
Biological: intravenous immunoglobulins — One course of Intravenous Immunoglobulins 0.4 g/kg/die for 5 consecutive days
  Arms: intravenous immunoglobulins
Biological: Saline solution — Placebo
  Arms: saline solution

SUMMARY:
Postpolio syndrome is a condition that affects many polio survivors years after the acute infection and causes symptoms to increase or new symptoms to develop. Proinflammatory cytokine production within the central nervous system (CNS) indicates an underlying inflammatory process, amenable to immunomodulatory therapy. In this study the investigators sought to confirm that antiinflammatory treatment with intravenous immunoglobulin improves the disease.

ELIGIBILITY:
Inclusion Criteria:

* a history of acute poliomyelitis
* increased muscle weakness, muscle fatigue and pain in muscle groups previously affected by poliomyelitis
* a diagnosis of postpolio syndrome according to the criteria of Halstead and Rossi

Exclusion Criteria:

* clinically relevant systemic disease
* malignancy
* hypothyroidism
* diabetes mellitus not fully controlled by medical therapy
* medical or orthopedic disorders that could give rise to symptoms mimicking post-polio syndrome
* conditions associated with prolonged coagulation time
* serum IgA deficiency
* previous allergic reaction to IVIG
* body-mass index greater than 30
* immune-modulating treatments other than IVIG within the preceding 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
SF-36 physical component | Baseline; 2 and 4 months after treatment